CLINICAL TRIAL: NCT00786227
Title: Initial Validation of PROMIS Physical Function/Disability Scales in Rheumatoid Arthritis (RA)
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); QualityMetrics (Industry)
Responsible Party: Sponsor
Other Study IDs: 07-01; 5U01AR052158 (NIH); 5U01AR052158-02 (NIH)
Record Dates: First submitted 2008-11-05; First posted 2008-11-06 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Legacy HAQ-DI first, PROMIS 20-item short form first: To eliminate effects due to order of administration, patients with RA will be randomized to complete either the Legacy measure HAQ-DI first in the assessment battery or the PROMIS 20-item short forms first.

SUMMARY:
The Patient-Reported Outcomes Measurement Information System (PROMIS) is an NIH Roadmap initiative to develop a computerized system measuring patient-reported outcomes in respondents with a wide range of chronic diseases and demographic characteristics. In the first four years of its existence, the PROMIS network developed item banks for measuring patient-reported outcomes in the areas of pain, fatigue, emotional distress, physical function, and social functioning. During the item banking process, the PROMIS network conducted focus groups, individual cognitive interviews, and lexile (reading level) analyses to refine the meaning, clarity, and literacy demands of all items. The item banks were administered to over 20,000 respondents and calibrated using models based on item response theory (IRT). Using these IRT calibrations, computerized adaptive test (CAT) algorithms were developed and implemented. The network has designed a series of studies using clinical populations to evaluate the item attributes, examine their utility as CATs, and validate the item banks. More information on the PROMIS network can be found at www.nihpromis.org.

DETAILED DESCRIPTION:
This is a longitudinal clinical validation study of the PROMIS physical function, fatigue, and pain impact short forms in patients with rheumatoid arthritis (RA). Patients will complete assessments at two points: baseline and 6 months post-baseline. The responsiveness of six PROMIS static forms (physical function [HAQ, PF-10, 10 and 20 item short forms], fatigue, and pain impact) will be evaluated for change over the 6-month period. Physical function change scores will be contrasted with established Legacy physical function instruments. The test of "responsiveness" is defined as the ability of the instrument to detect change after major treatment intensification, self-reported improvement in functioning, or positive changes in patient global scores. The order of presentation of forms will be randomly assigned to eliminate questionnaire fatigue or other order effects as factors. We will also evaluate the test-retest reliability of four PROMIS static forms (HAQ and PF-10 physical function, fatigue, and pain impact) in a random subsample of patients at 1-week post-baseline. In addition, we will evaluate convergent validity of PROMIS measures of physical function by comparing self-report with observation of performance of physical function tasks in a subsample of patients randomly selected from the local geographic region.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatologist-diagnosed RA
* Meets one of the conditions for treatment intensification as described in the protocol
* Ability to read, write, and speak English
* Ability to understand and provide informed consent

Exclusion Criteria:

* Unable or unwilling to complete questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from three sources will be included in the study: ARAMIS RA cohort, Stanford RA registry, and Stanford RA clinical trials patients.
Sampling Method: Probability Sample
Enrollment: 761 (Actual)
Dates: Start 2008-06; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Ability of Legacy or PROMIS instruments to detect change over 6 and 12 months in RA: (a) when an anti-TNF drug has been begun, (b) when the patient reports improvement over the prior period, (c) when the patient global has improved over the prior period | Measured at 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: James F. Fries, MD, Principal Investigator — Stanford School of Medicine
Locations (1):
- Stanford University School of Medicine, Palo Alto, California, United States